CLINICAL TRIAL: NCT01409746
Title: Early Brain Development in Twins
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 03-0989; R01MH070890-05 (NIH)
Record Dates: First submitted 2009-04-06; First posted 2011-08-04 (Estimated); Last update posted 2020-05-11 (Actual); Status verified 2020-03

CONDITIONS: Twin Brain Development
Keywords: twin; brain development; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — buccal swabs; MRIs, ultrasounds
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- twins: twin pairs

SUMMARY:
The purpose of this study is to study the role of genes and environment in early brain development using a twin approach. The investigators will use magnetic resonance imaging (MRI) to study brain structure and it's relationship to cognitive development. Specifically, the investigators will study cortical gray and white matter volumes, volumes of subcortical structures and cerebellum, as well as diffusion properties in major white matter tracts using DTI tractography.

DETAILED DESCRIPTION:
Twin studies have been critical in determining the contributions of genetic and environmental factors to normal brain structure and for understanding abnormalities of brain development that underlie neurodevelopmental and neuropsychiatric disorders. In adults and older children, twin studies indicate that genes play a significant role in the variability of global brain volumes, including total brain, total gray and total white matter volumes. Other than this current study, there have been no studies of twin brain development in early childhood, the period of brain development implicated in the pathogenesis of many psychiatric disorders. In the first funding cycle of this grant, the investigators used prenatal ultrasound and neonatal MRI to study discordance of early brain development, and to determine genetic and environmental contributions to neonatal brain structure. The investigators have and have developed a unique and valuable cohort of twins, having recruited and scanned over 100 twin pairs. The investigators found that discordance of prenatal brain size in MZ twins is similar to that in DZ twins, but that by 1 month after birth, discordance of overall brain volume in MZ twins is already less than in DZ twins. Contrary to our original hypothesis, statistical modeling of neonatal MRI brain volumes in our twin cohort indicates that global tissue volumes are highly heritable, similar to that observed in older children and adults. Therefore, it appears that genetic programs act very early in postnatal brain development to determine global tissue volumes. Interestingly, preliminary longitudinal mapping of correlations in gray matter density indicate correlations decrease in the first year of life, perhaps as the result of rapid brain growth in the first years of life. The investigators also found that while global white matter volumes are highly heritable, diffusion tensor properties of specific white matter tracts are not. In the next funding cycle, the investigators propose to continue enlarging this unique cohort and to follow them through age 6 years with structural MRI, diffusion tensor imaging (DTI), and developmental assessments to determine how genetic and environmental factors contribute to brain development in the first years of life.

ELIGIBILITY:
Inclusion Criteria:

* twins

Exclusion Criteria:

* major medical, obstetrical or neurological complications

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: medical center and community sample
Sampling Method: Non-Probability Sample
Enrollment: 550 (Actual)
Dates: Start 2004-04; Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Brain Gray Matter Volume | Change in heritability from birth to age 6 years
  Will assess gray matter volume with MRI and use structural equation modeling to determine relative contributions of genes and environment to variation of gray matter volumes.
Brain white matter tract integrity | Change in heritability from birth to age 6 years
  Will assess white matter tract development and integrity using diffusion tensor imaging and will determine relative contributions of genes and environment ot this using twin methodology.

SECONDARY OUTCOMES:
Mullen composite Score | 1,2,4,6 years
  Will assess genetic and environmental contributions to early cognitive development using a twin methodology

CONTACTS AND LOCATIONS:
Overall Officials: John H Gilmore, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- UNC Department of Psychiatry, Chapel Hill, North Carolina, United States

REFERENCES:
- [Result] Mukherjee N, Kang C, Wolfe HM, Hertzberg BS, Smith JK, Lin W, Gerig G, Hamer RM, Gilmore JH. Discordance of prenatal and neonatal brain development in twins. Early Hum Dev. 2009 Mar;85(3):171-5. doi: 10.1016/j.earlhumdev.2008.07.008. Epub 2008 Sep 19. PMID 18804925
- [Result] Gilmore JH, Schmitt JE, Knickmeyer RC, Smith JK, Lin W, Styner M, Gerig G, Neale MC. Genetic and environmental contributions to neonatal brain structure: A twin study. Hum Brain Mapp. 2010 Aug;31(8):1174-82. doi: 10.1002/hbm.20926. PMID 20063301
- [Result] Knickmeyer RC, Kang C, Woolson S, Smith JK, Hamer RM, Lin W, Gerig G, Styner M, Gilmore JH. Twin-singleton differences in neonatal brain structure. Twin Res Hum Genet. 2011 Jun;14(3):268-76. doi: 10.1375/twin.14.3.268. PMID 21623657
- [Result] Geng X, Prom-Wormley EC, Perez J, Kubarych T, Styner M, Lin W, Neale MC, Gilmore JH. White matter heritability using diffusion tensor imaging in neonatal brains. Twin Res Hum Genet. 2012 Jun;15(3):336-50. doi: 10.1017/thg.2012.14. PMID 22856369
- [Result] Li Y, Gilmore JH, Wang J, Styner M, Lin W, Zhu H. TwinMARM: two-stage multiscale adaptive regression methods for twin neuroimaging data. IEEE Trans Med Imaging. 2012 May;31(5):1100-12. doi: 10.1109/TMI.2012.2185830. Epub 2012 Jan 24. PMID 22287236
- [Result] Lee SJ, Steiner RJ, Luo S, Neale MC, Styner M, Zhu H, Gilmore JH. Quantitative tract-based white matter heritability in twin neonates. Neuroimage. 2015 May 1;111:123-35. doi: 10.1016/j.neuroimage.2015.02.021. Epub 2015 Feb 17. PMID 25700954
- [Result] Gao W, Elton A, Zhu H, Alcauter S, Smith JK, Gilmore JH, Lin W. Intersubject variability of and genetic effects on the brain's functional connectivity during infancy. J Neurosci. 2014 Aug 20;34(34):11288-96. doi: 10.1523/JNEUROSCI.5072-13.2014. PMID 25143609
- [Result] Jha SC, Xia K, Ahn M, Girault JB, Li G, Wang L, Shen D, Zou F, Zhu H, Styner M, Gilmore JH, Knickmeyer RC. Environmental Influences on Infant Cortical Thickness and Surface Area. Cereb Cortex. 2019 Mar 1;29(3):1139-1149. doi: 10.1093/cercor/bhy020. PMID 29420697
- [Result] Lee SJ, Zhang J, Neale MC, Styner M, Zhu H, Gilmore JH. Quantitative tract-based white matter heritability in 1- and 2-year-old twins. Hum Brain Mapp. 2019 Mar;40(4):1164-1173. doi: 10.1002/hbm.24436. Epub 2018 Oct 27. PMID 30368980
- [Result] Jha SC, Xia K, Schmitt JE, Ahn M, Girault JB, Murphy VA, Li G, Wang L, Shen D, Zou F, Zhu H, Styner M, Knickmeyer RC, Gilmore JH. Genetic influences on neonatal cortical thickness and surface area. Hum Brain Mapp. 2018 Dec;39(12):4998-5013. doi: 10.1002/hbm.24340. Epub 2018 Aug 24. PMID 30144223